CLINICAL TRIAL: NCT02311075
Title: Determination of the Mechanisms Involved in Conduit Artery Endothelial Dysfunction in Type 2 Diabetes
Brief Title: Mechanisms of Endothelial Dysfunction in Type 2 Diabetes
Acronym: DIAB-EETs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013/049/HP; 2013-A01107-38 (Other: ANSM)
Record Dates: First submitted 2014-11-25; First posted 2014-12-08 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patient comparative approach (Experimental): Assessing the availability of biological markers (NO, EETs, ET-1 and ROS) during endothelial stimulation using blood samples.
  Interventions: Biological: Blood samples
- Control subjects comparative approach (Experimental): Assessing the availability of biological markers (NO, EETs, ET-1 and ROS) during endothelial stimulation using blood samples.
  Interventions: Biological: Blood samples
- Healthy volunteers metabolic approach (Experimental): Assessing the availability of biological markers (NO, EETs, ET-1 and ROS) during endothelial stimulation using blood samples during hyperglycemia or hyperinsulinemia.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — Blood samples will be performed at baseline and during endothelial stimulation by hand skin heating to quantify metabolites of NO, EETs, ET-1 and ROS

SUMMARY:
Endothelial dysfunction of conduit arteries plays an important role in the development of cardiovascular complications associated with type 2 diabetes. In order to propose targeted therapeutic approaches, this study aim to determine the mechanisms involved in endothelial dysfunction of conduit arteries in these patients.

ELIGIBILITY:
Inclusion Criteria:

- Type 2 diabetic patients or control subjects or healthy volunteers

Exclusion Criteria:

* Macroangiopathy
* Insulin treatment
* Chronic kidney disease (eGFR<60 ml/min/m²)
* Hyperlipidemia (total cholesterol>2.5 g/l)
* Smoking habit > 5 cigarettes/day
* Pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in EET concentration during endothelial stimulation | 30 min from the beginning of hand skin heating

SECONDARY OUTCOMES:
Change from Baseline in NO concentration during endothelial stimulation | 30 min from the beginning of hand skin heating
Change from Baseline in ET-1 concentration during endothelial stimulation | 30 min from the beginning of hand skin heating
Change from Baseline in ROS concentration during endothelial stimulation | 30 min from the beginning of hand skin heating

CONTACTS AND LOCATIONS:
Overall Officials: Robinson JOANNIDES, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Derived] Duflot T, Moreau-Grange L, Roche C, Iacob M, Wils J, Remy-Jouet I, Cailleux AF, Leuillier M, Renet S, Li D, Morisseau C, Lamoureux F, Richard V, Prevost G, Joannides R, Bellien J. Altered bioavailability of epoxyeicosatrienoic acids is associated with conduit artery endothelial dysfunction in type 2 diabetic patients. Cardiovasc Diabetol. 2019 Mar 18;18(1):35. doi: 10.1186/s12933-019-0843-z. PMID 30885203